CLINICAL TRIAL: NCT00322699
Title: Sequential Whole Bladder Photodynamic Therapy (WBPDT) in the Management of Superficial Bladder Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: North Florida/South Georgia Veterans Health System (Other)
Collaborators: North Florida Foundation for Research and Education (Other); Axcan Pharma (Industry)
Responsible Party: Principal Investigator, Unyime O. Nseyo, MD, PHYSICIAN, North Florida/South Georgia Veterans Health System
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WBPDT-577-04
Record Dates: First submitted 2006-05-04; First posted 2006-05-08 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2011-08

CONDITIONS: Superficial Bladder Cancer
Keywords: Bladder Cancer; Photodynamic Therapy; Photofrin; Photosensitization; Photoradiation
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Urinary Bladder Neoplasms; Photosensitivity Disorders | interventions — Dihematoporphyrin Ether

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A single arm, non-randomized Phase II Study (Experimental): Non-Randomized Phase II,Single Arm Study evaluating the efficacy of whole bladder photodynamic therapy as an alternative to radical cystectomy.
  Interventions: Procedure: Whole bladder laser light treatment as an alternative to radical cystectomy; Drug: Photofrin

INTERVENTIONS:
Procedure: Whole bladder laser light treatment as an alternative to radical cystectomy — The drug,Photofrin,at the dose of 1.5 mg/kg is infused intravenously two days prior to performing whole bladder laser light (630 nm) treatment.
Drug: Photofrin — The drug,Photofrin,at the dose of 1.5 mg/kg is infused intravenously two days prior to performing whole bladder laser light (630 nm) treatment.
  Other Names: Porfimer Sodium, Photofrin,photosensiter,dye

SUMMARY:
This protocol is evaluating efficacy and toxicity of three sequential whole bladder photodynamic treatment with Photofrin and red laser light (630 nm) in the management of superficial bladder cancer (non-muscle invasive) in those patients who have failed or are not candidates for conventional intravesical therapy.

DETAILED DESCRIPTION:
Patient Evaluation and Treatment:

1. Patients will sign an IRB-approved informed consent form
2. Initial patient assessments will include:

   * eligibility
   * History and physical.
   * clinical profile
   * upper urinary tract imaging (if clinically indicated)
   * urinary symptoms assessment

WBPDT Treatment:

1. Porfimer Sodium (Photofrin) 1.5 mg/kg iv followed 2 days later by whole bladder laser light at 630 nm with target light doses of 1200 Joules (+/-100Joules)
2. Patients will undergo three sequential WBPDT treatments
3. Treatments will occur at least three months apart
4. All WBPDT treatments will occur within 12 months

   Decisions to administer a second or third WBPDT will be based upon urological and medical assessment of the individual patient and not necessarily dependent upon Dose Limiting Toxicities (DLT) or early stopping endpoints (although such information may be taken into account in the individual patient assessment). Patients experiencing DLT may continue WBPDT at the investigator's discretion at the same or reduced doses of Porfimer Sodium and/or light.

   The following will be considered Dose Limiting Toxicities (DLT):
   * Urinary symptoms grade 3, or more over 12 weeks duration (see section 7 for toxicity grading)
   * Loss of > 50% of baseline bladder volume
   * Clinical decision of investigator or patient to discontinue due to toxicity.

   Efficacy will be assessed on the basis of the following criteria:
   * Complete Response: cystoscopy with biopsy and/or cytology without evidence of cancer.
   * Partial Response: normal cystoscopy and biopsies, if obtained, but persistent positive or suspicious cytology localized to the bladder; or, for patients with CIS, > 50% reduction in extent of CIS.
   * Persistent/Recurrent Disease: persistent or recurrent cancer of the same or lesser stage and grade as at enrollment without obvious increase in tumor burden.
   * Progression: cancer of any greater stage or grade than at enrollment or obvious increase in tumor burden.

   Referred patients will undergo post-PDT cystoscopy by the referring Urologists, who will transmit the results to the study site in Gainesville,Fl.
5. Symptoms will be assessed for one month following each WBPDT by weekly telephone contact.
6. Urine and blood for cytokines will be obtained before each treatment and possibly twice afterwards and stored -80oF for analysis later.
7. Biopsy specimen samples from tumor and normal bladder may be obtained at cystoscopy and stored for later analysis for biomarkers.
8. Patients will be followed for toxicity, disease status, urinary tract symptoms, and survival.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of bladder cancer, non muscle invasive
* Recurrent after at least one course of standard intravesical therapy after transurethral resection (TURBT).
* Maximum debulking of tumor by TURBT/fulguration
* One or more of the following:

  * Contraindications to conventional intravesical therapy, including patient's refusal.
  * Positive or suspicious urine cytology localized to the bladder
  * Prior intravesical therapy and persistent atypia.
  * Premalignant (diffuse squamous metaplasia or malakoplakia) lesions.
* Bladder capacity greater or equal to 150 cc.
* No contraindications to an appropriate anesthesia or analgesia.
* Karnofsky's performance status > 50.
* Patients must sign an informed consent form in accordance with the Institution's Review Board and FDA 21 CFR Part 50.
* Female patients must be practicing a medically acceptable form of birth control or be sterile or postmenopausal.

Exclusion Criteria:

* Pregnant or nursing mother.
* Known hypersensitivity to porphyrins.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-02; Primary Completion 2010-04 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | 18 months

SECONDARY OUTCOMES:
Disease progression | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Unyime O Nseyo, M.D., Principal Investigator — NF/SGVAHS
Locations (1):
- Malcom Randall NF/SG Veterans Administration Health System, Gainesville, Florida, United States